CLINICAL TRIAL: NCT07201870
Title: A Pilot Feasibility Study of the Implementation, Usability, Acceptability and Effectiveness of an Online Bariatric Surgery Preparation Platform
Brief Title: Digital Preparation for Bariatric Surgery: Feasability Pilot Trial
Acronym: Pilot Be-Ready
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Sylvain Iceta, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-4306
Record Dates: First submitted 2025-08-06; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Bariatric Surgery Patients; Online Education; eHealth Literacy; Online-Intervention; Usability Satisfaction; Implementation Strategies; Shared Decision Making
Keywords: obesity; bariatric surgery; preparation; education platform
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The 3 arms will be evaluated at baseline, after 3 months and after 6 months. The control group (Arm 1) will then follow a sequential study model and follow the same course ass arm 3. This will ensure equality of car for every participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Control arm (No Intervention): Participants will follow the standard protocols of preparation for a bariatric surgery and remain on the waiting list without access to the educational platform (Precare). Participants will have to fulfill the participant's description module and the readiness assessment. After the 6-month assessment, the patient will be providing a full access to Precare and will follow the same assessment process as arm 3 (i.e., Precare usability module, and the secondary clinical assessment module).
- Arm 2: active arm with a short assessment (Experimental): Participants randomized to the active arm with a short assessment (arm 2) will be provided with 6-month of full access to the educational platform Precare and will have to fulfill the participant's description module and the readiness assessment (same as arm 1), as well as the Precare usability module.
  Interventions: Other: Acces to Precare online platform
- Arm 3: active arm with a full assessment (Experimental): Participants randomized to the active arm with a full assessment (arm 3) will be provided with 6-month of full access to the educational platform Precare after having fulfilled a REDCap module, including the participant's description module, the readiness assessment, the Precare usability module, and the secondary clinical assessment module.
  Interventions: Other: Acces to Precare online platform

INTERVENTIONS:
Other: Acces to Precare online platform — Precare is an online educational platform for patients on the waiting list for bariatric surgery. Precare offers personalized educational content as well as a calendar and appointment management system. It has been accredited by the Quebec Ministry of Health and Social Services.
  Arms: Arm 2: active arm with a short assessment; Arm 3: active arm with a full assessment

SUMMARY:
Metabolic and bariatric surgery (MBS) is in increasing demand due to the growing prevalence of severe obesity and the cumulating evidence of long-term benefits on weight loss, cardiometabolic and functional health outcomes, and quality of life for individuals living with severe obesity. The time spent on the waiting list for an MBS follow the same trend with an estimated waiting time of more than 18 months and rising. The lack of resources and multidisciplinary capabilities among MBS centers impacts the quality of care and outcomes, which greatly contributes to delayed surgery. In 2023, 31% of patients who had an initial appointment with the MBS nurse at the Quebec Heart and Lung Institute - Laval University(IUCPQ) did not proceed with the surgery due to fear, uncertainty, or timing issues. Additionally, 49% reported that their concerns (e.g., financial, home support) were not addressed before MBS. These data highlight the urgent need to implement strategies to optimize wait time and ensure that MBS preparation is tailored to patients' expectations. Telehealth has significantly impacted surgical preparation, including for MBS, by enhancing accessibility, reducing dropout rates, and maintaining clinical outcomes that are comparable to traditional in-person visits but it requires real-time multidisciplinary execution, limiting the applicability for MBS waiting list patients. An interesting complement to telehealth intervention is online education platforms which offer digital flexibility, a significant advantage over in-person session.

To date, most MBS online resources are fee-based or driven by commercial interests and lack of clinical evidence, which raises concerns about their efficacy and safety for users who are seeking reliable support during their MBS journey.

A free online education platform could optimize the time spent on the MBS waiting list by increasing patients' readiness for MBS, furnishing invaluable insights into the patient journey to MBS, and empowering individuals undergoing MBS. The IUCPQ is in the process of working on the care trajectory of patients with obesity. The Healthcare Direction and the Bariatric Surgery Clinic decided to use a platform called Precare. This platform offers personalized educational content as well as a calendar and appointment management system. It has been accredited by the Quebec Ministry of Health and Social Services. The present research focuses on the pilot testing the implementation and effectiveness of the PreCare solution for patients awaiting bariatric surgery at the IUCPQ.

The objectives of the research proposal are: 1) To assess the usability and acceptability of the Precare platform using a mixed design methodology; 2) To evaluate the logistical feasibility of using the platform in a clinical setting; 3) To determine whether extensive self-questionnaire assessments may impact the use of the Precare platform; 4) To explore barriers and facilitators to enhance patient engagement and knowledge retention; and 5) To derive estimates variables related to gender, ethnicity, cultural background, learners and psychological profiles for future phases.

Our hypotheses are:

1. The Precare platform will exhibit high usability and acceptability.
2. Testing the Precare platform in real clinical settings is viable and will yield promising results for improving patient readiness for Metabolic and Bariatric Surgery.

ELIGIBILITY:
Inclusion Criteria:

* Be on the waiting list for metabolic and bariatric surgery at IUCPQ
* not yet assessed by the local team and with an expected wait time of more than 6 months
* understand French
* Have an active email address

Exclusion Criteria:

* Be part of the same household as someone already involved in this research project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Self-perceived barriers to metabolic and bariatric surgery | At baseline
  Short questionnaire to assess the barriers to the decision for bariatric surgery perceived by patients based on Luck-Sikorski C, Jung F, Dietrich A, Stroh C, Riedel-Heller SG. Perceived Barriers in the Decision for Bariatric and Metabolic Surgery: Results from a Representative Study in Germany. Obes Surg. 2019 Dec;29(12):3928-3936. doi: 10.1007/s11695-019-04082-1. PMID: 31301032.
eHeals Literacy Scale | At baseline
  Survey to measure Participants' feelings about their use of the Internet as a tool for obtaining health-related information. We will use the validated french version of the eHeals scale, a 10-item questionnaire. Question's response is measured with a 5 point likert scale with response options either going from 'strongle disagree' to 'strogly agree', 'not at all; usefull' to 'very usefull' or ' Not at all important' to 'Very important'. Higher scores represent higher sefl-perceive eHeals literacy.
Index of Learning Styles | At baseline
  To assess of the learner profile of the patient (44 items) Adapted from the Index of Learning Styles Questionnaire by Barbara A. Solomon & Richard M. Felder University of North Carolina Raleigh, NC 27695
University of Rhode Island Change Assessment Scale (URICA) | At baseline, 3 months and 6 months
  32-item scale based on Prochaska and DiClemente's transtheoretical behaviour change model to assess the readiness of the patient to bariatric surgery. Each question is measured on a 5-point Likert scale with response options ranging from "strongly disagree"(1 point) to "strongly agree"(5 points). Questions are divided into four subscales of 8 items each: precontemplation, contemplation, action and maintenance. Each subscale score from 1 to 40. The readiness to bariatric surgery score is calculated by adding the scores from the Contemplation, Action and Maintenance subscales and subtracting from that sum the Precontemplation subscale score. The total score ranges from 1 to 160, with higher scores indicating better readiness.
Home-made survey | At baseline, 3 months and 6 months
  To assess readiness of the patient to bariatric surgery. Questionnaire based on the current questionnaire sent to participants when they attempt psychiatric assessment for metabolic and bariatric surgery at the Quebec Heart and Lung Institute - Laval University(IUCPQ)
System Usability Scale score(SUS) | at 3 and 6 months
  To asses the usability of the platform Precare based. SUS is a 10-item validated questionnaire for assessing system usability, including software, websites, and applications. Each item is rated on a 5 points Likert scale ranging from 'Strongly disagree'(1) to 'strongly agree'(5). A higher score represent a higher usability of the platform. (only for arm 2 and arm 3)

SECONDARY OUTCOMES:
Mental Health Continuum Short Form | At baseline, 3 months and 6 months
  14-item questionnaire to assess overall psychopathology. Each question is measured on a 6-point Likert scale with response options ranging from "Never"(0 point) to "Everyday"(5 points). Total score ranges from 0 to 70, with a higher score representing better mental well-being. (Only for arm 3)
Motivation to attempt metabolic and bariatric surgery | At baseline
  Survey on factors influencing patients' mottivation to undergo bariatric surgery
Physical and psychological comorbidities | At baseline
  Number of current associated comorbidities to patient
Body Mass Index in kg.m-2 | At baseline
  Anthropometric markers: weight and height will be combined to report the body mass index (BMI) in kg/m^2
Age of first weight gain | At baseline
  Age of participants when they first gained weight
Weight Loss Attempts | At Baseline
  Description of past weight loss attempts as reported by participant
Adherence to weight loss attempts | At baseline
  Duration of adherence to the various approaches of weight loss tried by participants
Minimal weight | At baseline
  Minimum weight reached by the participant since adulthood
Maximum weight | At baseline
  Maximum weight reached by the participant since adulthood
Binge Eating Scale score | At baseline, 3 months and 6 months
  To assess the presence of certain binge eating behaviors that may be indicative of an eating disorder. The higher the score, the more binge eating behaviors is observed. The minimum score is 0 while the maximum score is 46. The final result allows to say if the person has an absent (less than 17), moderate (between 18 and 26) or severe (more than 27) binging level. (Only for arm 3)
modified Yale Food Addiction Scale 2.0 (mYFAS 2.0) | At baseline, 3 months and 6 months
  The mYFAS 2.0 was designed to assess food addiction using a shorter version than the YFAS 2.0.It assesses the symptoms of food addiction and the resulting distress and impaired functioning. The higher the level of symptoms, the more severe the food addiction. Impaired functioning and distress are scored from 0 to 2. Symptoms are scored from 0 to 11. If the functioning and distress score is 1 and above, the food addiction may be mild (2-3 symptoms), moderate (4-5 symptoms), or severe (6+ symptoms). (Only for arm 3)
Hospital Anxiety and Depression Scale (HADS) | At baseline, 3 months and 6 months
  This self-administered questionnaire assesses depressive symptoms using seven items (ÉHAD-D) and anxiety symptoms using another seven items (ÉHAD-A), for a total of 14 items. Each question is scored from 0 to 3. Higher scores indicate higher level of anxiety and depression. A total score between 0 and 7 reflects a normal level of anxiety and depression, a score of 8 to 10 indicates a borderline level and a score of 11 and above indicates a high level of anxiety and depression. (Only for arm 3)
Canadian Food Intake Screener | At baseline, 3 months and 6 months
  To assess the participant's degree of adherence to the Canada's food guide (Only for arm 3)
Canadian Eating Practices Screener | At baseline, 3 months and 6 months
  To assess the participant's degree of adherence to the Canada's food guide (Only for arm 3)
Malnutrition Screening Tool | At baseline, 3 months and 6 months
  To assess participant's risk of malnutrition scored from 0 to 7. A score of 2 or more means the participant is at risk for malnutrition. (Only for arm 3)
Global Physical Activity Questionnaire | At baseline, 3 months and 6 months
  Questionnaire from the World Health Organization to assess physical activity participation of the patient (Only for arm 3)
Multidimensional Body Self Relations Questionnaire-Appearance Scales | At baseline, 3 months and 6 months
  34-item questionnaire to assess aspects of body image. Questions are divided into five subscales: Appearance Evaluation, Appearance Orientation, Body Area Satisfaction, Overweight Preoccupation and Self-classified Weight. Each question is measured with 5-point Likert scales. The mean of each subscale is calculated. Higher scores generally indicate more positive body image and appearance satisfaction (Only for arm 3)
Multidimensional Scale of Perceived Social Support | At baseline, 3 months and 6 months
  12-Item questionnaire to assess the social support of patients. Each question is measured on a 7-point Likert scale with response options ranging from " very strongly disagree"(1 point) to "very strongly agree"(7 points). Questions are divided into three subscales of four items each: Significant others, Friends and Family. Each subscale score ranges from 4 to 28. A higher score indicates a higher perceived support. (Only for arm 3)
World Health Organization Quality of Life- BREF | Art baseline, 3 mopnths and 6 months
  26-item questionnaire to assess the quality of life of the patient. Each question is measured on 5-point Likert scales. Total score ranges from 0 to 100, with higher score associated to better quality of life. (Only for arm 3)
Patient Empowerment Strategies Questionnaire | At baseline, 3 months and 6 months
  15-item questionnaire to assess the patient empowerment. Each question is measured on a 4-point Likert scale with response options ranging from "totally agree"(4 point) to "totally disagree"(1 points). Score ranges from 15 to 54. Higher scores indicate greater patient empowerment. (Only for arm 3)
Recruitment rate | Through study completion, an average of 2 year
  Assessed by calculating the ratio of participants recruited for the current study / number of participants invited to participate in the present study.
Recrutement time | Through study completion, an average of 2 year
  Assessment of the time needed to recruit the current study population
Time before first connection | Through study completion, an average of 2 year
  Assessment of the time between logging sent and the first connection
Retention rate | Through study completion, an average of 2 year
  Assessement of the pourcentage of participants who finish every steps of the study
missing and incongruent data | Through study completion, an average of 2 year
  Percentage of missing and incongruent data
Time to complete the initial assessment | Through study completion, an average of 2 year
  Assessment of the mean time to complete the initial assessment (overall and per questionnaires)
Response time per questionnaire | Through study completion, an average of 2 year
  The participant's time to answer each questionnaire
Questionnaires reliability index | Through study completion, an average of 2 year
  the congruence of questionnaires reliability index with the literature
website performance indicators | Through study completion, an average of 2 year
  Assessment of the time to request and compute website performance indicators
Participant's learner profile. | Through study completion, an average of 2 year
  The percentage of users classified in a learner profile.
Active User Rate | At 3 and 6 months
  Percentage of registered users who are actively using the platform
Session duration | At 3 and 6 months
  Average amount of time users spend on the platform per session
Views per session | At 3 and 6 months
  Number of pages views per session
Login frequency | At 3 and 6 months
  Participant's login frequency
Completion rates | At 3 and 6 months
  Completion rate for each module of the platform PreCare
Bounce rate | At 3 and 6 months
  Percentage of visitors who navigate away from the site after viewing only one page
Participants' Pathways | At 3 and 6 months
  Assessment of the pathways followed by users (individual and cluster analysis), viewing and download rates
Content revisit rate | At 3 and 6 months
  Number of time users come back to a page
Platform uptime | At 3 and 6 months
  Tracking of the PreCare platform's uptime; time the platform has been operationnal during the study
Platform load times | At 3 and 6 months
  Tracking the PreCare platform's load time ; time it take the platform to display the requested page
Platform's error rates | At 3 and 6 months
  Tracking the PreCare platform's error rates; number of error occuring

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ, Québec, Quebec, Canada